CLINICAL TRIAL: NCT00556075
Title: A Phase II, Three-Arm, Parallel Design, Dose-Ranging Placebo-Controlled, Randomized, Double-Blind, Multicenter Study Evaluating the Safety and Efficacy of Proellex in the Treatment of Premenopausal Women With Symptomatic Endometriosis
Brief Title: Safety and Efficacy Study to Evaluate Proellex in the Treatment of Premenopausal Women With Symptomatic Endometriosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical hold for safety
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZPE-201
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pelvic pain; Oral progesterone blocker
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo
- 25 mg (Experimental): Proellex 25 mg once daily
  Interventions: Drug: Proellex 25 mg
- 50 mg (Experimental): Proellex 50 mg once daily
  Interventions: Drug: Proellex 50 mg

INTERVENTIONS:
Drug: Proellex 25 mg — 1 capsule daily for 4 months
  Arms: 25 mg
Drug: Placebo — 1 capsule daily for 4 months
  Arms: Placebo
Drug: Proellex 50 mg — 2 capsules daily for 4 months
  Arms: 50 mg

SUMMARY:
The purpose of this study is to determine whether Proellex is safe and effective for the treatment of symptomatic endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 18-48 inclusive
* Endometriosis documented by laparoscopic or surgical assessment within the past ten (10) years
* Clinical symptoms of endometriosis for at least the past three (3) months
* Endometriosis symptoms
* Must be sexually active unless sexually inactive for endometriosis-related dyspareunia
* Must have a regular or steady menstrual cycle lasting from 24 to 36 days and a detectable ovulation during the baseline period using an ovulation monitoring kit (for timing of endometrial biopsy)
* Other inclusion criteria may apply

Exclusion Criteria:

* Six (6) months or more without a menstrual period, or
* Prior hysterectomy or
* Prior bilateral oophorectomy
* Diagnosis of osteopenia
* Present history or condition that causes non-endometriosis-related dyspareunia
* Presence of excessive bleeding or menorrhagia
* Abnormal screening endometrial biopsy
* Other exclusion criteria may apply

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre vanAs, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (17):
- United States (17):
  - Advanced Clinical Therapeutics, LLC, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Medical Center for Clinical Research, San Diego, California
  - Compass Clinical Research, San Ramon, California
  - Altus Research, Lake Worth, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Medical Associates, Dubuque, Iowa
  - Physicians for Women, Cary, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - HWC Women's Research Center, Miamisburg, Ohio
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Gaffney Pharmaceutical Research, Gaffney, South Carolina
  - Greenville Pharma Research, Greenville, South Carolina
  - Advanced Research Associates, Corpus Christi, Texas
  - Clinical Trials of Texas/Institute for Women's Health, San Antonio, Texas
  - Clinical Trials of Texas/Seven Oaks Women's Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- C Placebo: Placebo: 1 capsule daily for 4 months
- A 25 mg: Proellex 25 mg: 1 capsule daily for 4 months
- B 50 mg: Proellex 50 mg: 2 capsules daily for 4 months
Period: Overall Study
Arm/Group | C Placebo | A 25 mg | B 50 mg
Started | 22 | 22 | 23
Completed | 9 | 13 | 15
Not Completed | 13 | 9 | 8
Not completed — Lost to Follow-up | 3 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Protocol Violation | 1 | 1 | 3
Not completed — Not eligible | 1 | 1 | 2
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Personal issues | 4 | 1 | 0
Not completed — Endometrial stripe not viewed on 2 tvu | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 25 mg | 50 mg | Total
Number analyzed (Participants) | 22 | 22 | 23 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 23 | 67
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 23 | 67
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 23 | 67

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the 50 mg Proellex Group and Placebo Group in the Month 4 Subject Diary Composite Pain Score
Time Frame: 4 months
Population: Zero participants were analyzed because no data were collected due to early termination
Arm/Group | Placebo | 25 mg | 50 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Difference Between the 25 mg and 50 mg Proellex Groups and Placebo Group in the Month 4 Subject Diary Composite Pain Score
Time Frame: 4 months
Population: Zero participants were analyzed because no data were collected due to early termination
Arm/Group | Placebo | 25 mg | 50 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Difference Between Each Treatment Group in the Subject Diary Composite Pain Score at the Monthly Visits
Time Frame: monthly
Population: Zero participants were analyzed because no data were collected due to early termination
Groups:
- Placebo: Placebo: 1capsule daily for 4 months
- 25 mg: Proellex 25 mg
  Proellex 25 mg: 1 capsule daily for 4 months
- 50 mg: Proellex 50 mg
  Proellex 50 mg: 2 capsules daily for 4 months
Arm/Group | Placebo | 25 mg | 50 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time to Pain-free Assessments Using the Composite Pain Score as Determined by Data Recorded in the Subject Diaries
Time Frame: days
Population: Zero participants were analyzed because no data were collected due to early termination
Groups:
- Placebo: Placebo
  Placebo: 1 capsule daily for 4 months
Arm/Group | Placebo | 25 mg | 50 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Duration of Pain-free Assessments Using the Composite Pain Score as Determined by Data Recorded in the Subject Diaries
Time Frame: days
Population: Zero participants were analyzed because no data were collected due to early termination
Arm/Group | Placebo | 25 mg | 50 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: The Number of Days With Pain as Determined by Data Recorded in the Subject Diaries, Analyzed Between Treatment Groups at the Monthly Visits
Time Frame: days
Population: Zero participants were analyzed because no data were collected due to early termination
Arm/Group | Placebo | 25 mg | 50 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | 25 mg | 50 mg
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22 | 1/23
Other Adverse Events (participants affected / at risk) | 18/22 | 22/22 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | 25 mg (N=22) | 50 mg (N=23)
Elevated LFTs (Investigations) | 0 (0) | 0 (0) | 1 (1) — Subject taking 50 mg/day
Grand Mal Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Subject taking placebo. Attributed to water intoxication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | 25 mg (N=22) | 50 mg (N=23)
Adominal pain (Gastrointestinal disorders) | 5 | 3 | 8
Nausea (Gastrointestinal disorders) | 3 | 8 | 11
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1
Fatigue (General disorders) | 0 | 2 | 1
Irritability (General disorders) | 0 | 0 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 4 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 0
URI (Infections and infestations) | 4 | 1 | 4
UTI (Infections and infestations) | 1 | 3 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 3
Bone density decreased (Investigations) | 2 | 4 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 4
Headache (Nervous system disorders) | 1 | 4 | 6
Migraine (Nervous system disorders) | 0 | 0 | 2
Cervical cyst (Reproductive system and breast disorders) | 1 | 1 | 2
Endometrial disorder (Reproductive system and breast disorders) | 0 | 2 | 3
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 1 | 3
Ovarian cyst (Reproductive system and breast disorders) | 16 | 10 | 15
Parovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 4 | 7

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with complete study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights